CLINICAL TRIAL: NCT03028571
Title: Acute Sympathetic Blockade and Endogenous Glucose Production
Brief Title: Autonomic Blockade and Endogenous Glucose Production
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The investigators decided not to perform the study. No participants have been enrolled.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 150466
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Trimethaphan; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects will be studied twice, randomly assigned to star on the intact day (saline) or the blocked day (trimethaphan) and after 1 month cross to the other arm
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intact Day (Placebo Comparator): The rates of endogenous glucose appearance (Ra) and peripheral glucose uptake (Rd) will be measured during a regular insulin clamp with concomitant infusion of saline at 48 ml/hr IV
  Interventions: Other: Saline
- Blocked Day (Experimental): The rates of endogenous glucose appearance (Ra) and peripheral glucose uptake (Rd) will be measured during a regular insulin clamp with concomitant infusion of trimethaphan (4mg/min) IV.
  Interventions: Drug: Trimethaphan

INTERVENTIONS:
Drug: Trimethaphan — Trimethaphan 4 mg/min IV will be given as a pharmacological tool to study the role of the autonomic nervous system on the regulation of endogenous glucose production by the liver.
  Arms: Blocked Day
Other: Saline — IV saline at a rate of 48 mL/hr, will be given during the insulin clamp to resemble the volume infused in the intact day
  Arms: Intact Day

SUMMARY:
The investigators will test the null hypothesis that there will be no changes in the insulin-mediated suppression of endogenous glucose production (EGP) in response to autonomic blockade. To test this hypothesis, the investigators propose to determine the role of the autonomic nervous system in hepatic insulin resistance.

DETAILED DESCRIPTION:
In this study, the investigators will test the null hypothesis that there will be no changes in the insulin-mediated suppression of endogenous glucose production (EGP) in response to autonomic blockade. The investigators will measure EGP at baseline (EGPBsl) and during the last 30 minutes of a hyperinsulinemic euglycemic clamp (EGPClamp) on two different occasions (intact and Blocked study days). A double blinded randomize cross-over design will be used. Subjects will be randomized to either the intact or blocked days and a month later will be crossed-over to the other arm. The investigator performing the analysis will also be blinded to the treatments received. At baseline in both study days it is expected to see any differences since the same subject will serve as his own control. During the clamp, insulin suppresses EGP. In obese insulin resistant subjects this suppression should be blunted. If the hypothesis is correct, it is expected an improvement in the suppression by insulin of EGP during autonomic blockade only. For this study, the primary endpoint therefore, will be the EGP during the clamp between the intact and blocked days.

H0= {(EGPClamp)Blocked - (EGPClamp)Intact}=0]

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 and 60 years of age
* Hypertension defined by two or more properly measured seated blood pressure readings >130/85 mmHg or currently on antihypertensive medication. This will allow us to include subjects with "pre-hypertension."
* Obesity will be defined as having a body mass index (BMI) ≥ 30 kg/m2.
* Insulin resistance will be defined as a HOMA2 IR index ≥1.6
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Current smokers or history of heavy smoking (>2 packs/day)
* History of alcohol or drug abuse
* Previous allergic reaction to study medications
* Evidence of type I or type II diabetes (i.e. fasting glucose >126 mg/dl, use of anti-diabetic medications)
* Cardiovascular disease other than hypertension such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
* History of serious cerebrovascular disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Impaired renal function
* Anemia
* Treatment with phosphodiesterase 5 inhibitors
* Treatment with anticoagulants
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1 month preceding the study
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol (i.e., clinically significant abnormalities on clinical, mental examination or laboratory testing or inability to comply with protocol, inability to find IV access)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Endogenous Glucose Production | Duration of the study (4 hours)
  Amount of label glucose appearance

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States